CLINICAL TRIAL: NCT04034823
Title: KN035, a Single Domain PD-L1 Subcutanuous Injection Antibody, in Combination With Trastuzumab and Docetaxel in HER2-positive Breast Cancer
Brief Title: KN035 in Combination With Trastuzumab and Docetaxel in HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, JZhao, Doctor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN035-TH-HER2
Record Dates: First submitted 2019-07-25; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive breast cancer; PD-L1 immune checkpoint
MeSH Terms: interventions — envafolimab; Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN035 in combination with trastuzumab and docetaxel (Experimental)
  Interventions: Biological: KN035; Biological: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Biological: KN035 — KN035 5 mg/kg s.c. Q3W
Biological: Trastuzumab — 8 mg/kg IV loading followed by 6 mg/kg Q3W IV
Drug: Docetaxel — 100 mg/m2 Q3W IV

SUMMARY:
This is an open-label, single arm phase II trial to evaluate the efficacy, safety and tolerability of KN035 in combination with trastuzumab and docetaxel. Eligible patient will be enrolled and receive protocol defined therapies until progressive disease, unacceptable toxicity or withdrawal of informed consent. Tumor assessment will be performed according to RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female subjects with age 18 to 70 (inclusive) years at the time of consent
* LVEF ≥50% at baseline
* ECOG performance status of 0-1
* Have not received 1L treatment for recurrent or metastatic breast cancer
* Adequate organ function

Exclusion Criteria:

* History of exposure to the cumulative doses of doxorubicin > 400 mg / m2 or equivalent
* History of autoimmune diseases
* Active brain metastasis
* Concurrent diseases that compromise patient's safety

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response | 12 months
  To estimate the overall response rate (CR + PR) of KN035 in combination with trastuzumab and docetaxel in patients with recurrent or metastatic HER2-positive breast cancer.
  • Overall Response rate will include confirmed complete response (CR) + confirmed partial response (PR), as determined as per RECIST v1.1 criteria and assessed by the local investigator

SECONDARY OUTCOMES:
Adverse events | 12 months
  To characterize the toxicity of KN035 in combination with trastuzumab and docetaxel as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE)

OTHER OUTCOMES:
Disease control rate | 12 months
  To estimate the disease control rate (CR + PR + SD) of KN046 in combination with trastuzumab and docetaxel. Disease control rate will include complete response (CR], partial response (PR), and stable disease (SD), as per RECIST v1.1 criteria